CLINICAL TRIAL: NCT04197921
Title: A Feasibility Clinical Trial of Exablate for Low Intensity Focused Ultrasound Neuromodulation in Patients With Opioid Use Disorder (OUD) and/or Other Substance Abuse Disorders (SUDs)
Brief Title: Exablate for LIFU Neuromodulation in Patients With Opioid Use Disorder (OUD) and/or Other Substance Use Disorders (SUDs)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OUD001
Record Dates: First submitted 2019-12-09; First posted 2019-12-13 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-01

CONDITIONS: Opioid-use Disorder; Substance Use Disorders
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Sham/Active ExAblate Treatment Stage 1 and 2 (Other): Subject will undergo both Treatment 1 (sham) and Treatment 2 (with enhanced intensity). Subjects are blinded to the order of the sham vs active treatment.
  Interventions: Device: Exablate Model 4000 Type 2.0/2.1

INTERVENTIONS:
Device: Exablate Model 4000 Type 2.0/2.1 — There are two treatment stages. In both stages, the subject will receive both the sham and active ExAblate treatment, and be evaluated for 90 days post-treatment for adverse events. During Stage 1 the subject will receive the moderate intensity Exablate LIFU procedure. During Stage2, the subject will receive the enhanced intensity ExAblate LIFU procedure. The subjects are blinded as to the order of the sham vs active treatment.

SUMMARY:
The purpose of this clinical trial is to investigate Low Intensity Focused Ultrasound (LIFU) using the Exablate® Model 4000 Type 2.0/2.1 as an adjunctive neuromodulatory treatment for OUD (Opioid Use Disorder) and/or other Substance Use Disorders (SUDs) by assessing its safety and tolerability in subjects with OUD.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant females, age 18 - 60 years old
2. Subject meets DSM-5 criteria for OUD and/or other SUDs including alcohol (assessed via the SCID-5) of at least two years duration
3. Subject is currently receiving outpatient treatment from the WVU Comprehensive Opioid Addiction Treatment Program (COAT), Intensive Outpatient Program (IOP) or any other program which implements the COAT model; residential or inpatient treatment from the WVU Center for Hope and Healing or an affiliated WVU hospital; or receiving outpatient/inpatient/residential treatment from similar programs that are well known to the research team. If the subject is prescribed medication for AUD or OUD (e.g. buprenorphine-naloxone, naltrexone), they will be on a stable dose of the medication for the 7 days prior to the procedure. Stable is defined as within the therapeutic range but does not require same exact dose for 7 days.
4. Subject has been off opioids and other illicit substances, except for cannabis, confirmed via urine toxicology screen
5. The NAc is apparent on MRI such that treatment targeting can be performed directly (visible on MRI) and indirectly (using other anatomical structures for measurements)
6. Subject is able to communicate sensations during the Exablate Transcranial procedure
7. Subject is willing to cooperate with the study requirements including compliance with the regimen and completion of all study visits
8. Subject is able to make own medical decisions as determined by the clinical team
9. Subject has signed and received a copy of the approved informed consent form

Exclusion Criteria:

1. Subjects who are taking medications which may adversely interact with MOUD (See Appendix B for full list). Being on one of these medications would not automatically exclude a participant from study participation, does not automatically exclude a prospective subject from study participation. If a prospective or current subject is taking any medication listed in Appendix B, the study investigator is responsible for determining whether the subject is eligible for inclusion or continued study participation."
2. Subject with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices
3. Subject with known intolerance or allergies to the MRI contrast agent gadolinium (GADOVIST®)
4. Subject who are unable or unwilling to tolerate the required prolonged stationary position during treatment (approximately 2-3 hours)
5. More than 30% of the skull area traversed by the sonication pathway is covered by scars, scalp disorders (e.g., eczema), or atrophy of the scalp
6. Subject with implanted objects in the skull or the brain
7. Subject diagnosed with advanced kidney disease or on dialysis
8. Subject with impaired renal function with estimated glomerular filtration rate <30 mL/min/1.73m2
9. Subject with known unstable cardiac status or severe hypertension including:

   1. Documented myocardial infarction within six months of enrollment
   2. Unstable angina on medication
   3. Unstable or worsening congestive heart failure
   4. Left ventricular ejection fraction below the lower limit of normal
   5. History of a hemodynamically unstable cardiac arrhythmia
   6. Cardiac pacemaker
   7. Severe hypertension (diastolic BP > 100 on medication)
10. Subject with history of abnormal bleeding, hemorrhage, or coagulopathy
11. Subject receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage (e.g. Avastin) within one month of focused ultrasound procedure
12. Abnormal coagulation profile (PLT < 100,000/μl), PT (>13.9 sec) or PTT (>37.5 sec), and INR > 1.2. If values are outside the range of normal limits, any clinically significant value may be excluded as determined by a study investigator.
13. Subject with cerebrovascular disease as determined by MRI according to the Fazekas criteria. Grades II and III on the Fazekas scale should be excluded
14. Past or present diagnosis of schizophrenia, psychotic disorder, bipolar disorder, or untreated depression other than one determined to be substance induced (assessed via SCID-5)
15. Score of greater than 17 on the Hamilton Depression Rating Scale (HAM-D) or increased risk of suicide based on any positive response regarding passive or active suicidal ideation with or without intent over the past 3 months or lifetime history of active suicidal ideation with intent on the Columbia-Suicide Severity Rating Scale (C-SSRS) at baseline
16. History of suicide attempt
17. Parental history of completed suicide
18. Subject meet the criteria for Cluster A or B Personality Disorders (assessed via SCID-5-PD)
19. Diagnosis of dementia or any other disorder which has led to a clinically significant cognitive impairment (assessed via NIHTB-CB)
20. Subject with brain tumors
21. Subject with chronic pulmonary disorders e.g. severe emphysema, pulmonary vasculitis, or other causes of reduced pulmonary vascular cross-sectional area
22. Any known CNS infection or infection with the Human Immunodeficiency Virus (HIV) or Hepatitis C (HCV). A diagnosis of Hepatitis C (HCV) alone is not exclusionary as long as hepatic function laboratory values are deemed not clinically significant by a study investigator and are ≤ 1.5 times the upper limit of normal.
23. Subject who has had deep brain stimulation or a prior stereotactic ablation of the NAc, basal ganglia or thalamus
24. Subject who has been administered botulinum toxins into the arm, neck, or face for 5 months prior to baseline
25. Subject who is currently participating in another clinical investigation with an active treatment arm
26. Subject unwilling to abstain from illicit substance use during the course of the study
27. Subject is considered to be a poor surgical or study candidate, which may include, but is not limited to the following: any medical, social, or psychological problem that could complicate the required procedures and evaluations of the study in the judgment of the investigator
28. Subject is non-English speaking
29. Subject is pregnant or planning to be pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Estimated)
Dates: Start 2019-11-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Treatment Emergent Adverse Events | Post-ExAblate Procedure through 4 Month Follow-Up
  Safety will be assessed by recording all adverse events that are treatment related. Each Adverse Event will be documented for patterns of occurence.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Tampa General Hospital, Tampa, Florida
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Weill Cornell Medicine, New York, New York
  - West Virginia University: Rockefeller Neuroscience Institute, Morgantown, West Virginia

REFERENCES:
- [Derived] Mahoney JJ, Thompson-Lake DGY, Ranjan M, Marton JL, Carpenter JS, D'Haese PF, Arsiwala T, Suffridge J, Farmer DL, Finomore VS, Tirumalai P, Hodder SL, Rezai AR. A case report of focused ultrasound neuromodulation of the bilateral nucleus accumbens for methamphetamine use disorder. Exp Clin Psychopharmacol. 2025 Sep 1. doi: 10.1037/pha0000793. Online ahead of print. PMID 40892597